CLINICAL TRIAL: NCT05982964
Title: Impact of Scapula Position on Functionality and Balance in People With Chronic Low Back Pain
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Other Study IDs: E-85646034-604.02.02-62452
Record Dates: First submitted 2023-07-31; First posted 2023-08-09 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- back pain group
- Healthy volunteers

SUMMARY:
Chronic low back pain is defined as pain that lasts for more than 3 months or exceeds the expected recovery time.

DETAILED DESCRIPTION:
Chronic low back pain is defined as pain that lasts for more than 3 months or exceeds the expected recovery time.

ELIGIBILITY:
Inclusion criteria:

* Individuals between the ages of 18-65
* Individuals with low back pain for at least 3 months for the first group
* Not undergoing surgery related to the lumbar region
* Cases without lumbar steroid injection in the last 3 months
* Not having visual and hearing loss
* Having low back pain
* Cases without neurological problems
* Cases without tumor and infection in the lumbar region
* Exclusion criteria:
* Individuals under the age of 18
* Individuals with low back pain for less than 3 months for the first group
* Not having a musculoskeletal or neuromuscular disease that limits mobility,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our study was carried out on healthy and non-specific low back pain individuals who came to Bahçeşehir University.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold Algometer | 1 day
  The pressure algometer is a tool used to assess the pain threshold. The algometer used in this study is connected to a dial measuring the pressure in kilograms and pounds, and consists of a metal piston with a diameter of 1 centimeter at the tip, the smallest gap of which is 100 gr and 10 kg/cm².
Examining the Scapular Position | 1 day
  The lateral scapular glide test was used to evaluate the scapula position. In the first position, the arms were relaxed at the sides, the shoulder was in the neutral position, in the second position the patient's hands were positioned around the waist and the humerus was brought to medial rotation and abduction of 45 degrees, and in the third position, the humerus was placed in maximal medial rotation and 90-degree abduction.
Evaluation of Balance | 1 day
  The static and dynamic postural stability of all individuals included in the study were evaluated with the Biodex Balance System (BDS).
  For dynamic stability measurement, a total of 3 tests were conducted, with the platform in dynamic position, with each period lasting 20 seconds, giving the participant a rest period of 10 seconds in between. Afterwards, the average of these 3 tests was obtained automatically by the device. In the results obtained, it is possible to interpret that as the score approaches 0, the balance is maintained, and as it moves away from 0, the balance is deteriorated.
Proprioception Evaluation | 1 day
  An inclinometer is an instrument that records angular movements with respect to gravity. The inclinometer has many advantages such as precise measurement, digital display, and ease of use.
  In our study, inclinometer was used in the evaluation of proprioception. Measurements will be recorded in degrees.
Evaluation of Functionality | 1 day
  The Oswestry Low Back Pain Disability Questionnaire (OBAEA) was used to examine functionality in patients with chronic low back pain. This survey consists of 10 questions in total. Each question has 6 options and ranges from 0 to 5. Participants are asked to mark the option that best fits their individual situation. While 50 is the highest score, it is evaluated as mild functional disability between 1 and 10 points, moderate functional disability between 11 and 30 points, and severe functional disability between 31 and 50 points.
Waist Awareness Assessment | 1 day
  Fremantle Waist Awareness Questionnaire was used to evaluate low back awareness in the study. The Fremantle Waist Awareness Questionnaire is the only one that assesses body awareness about the waist. It consists of 9 questions in total and each question has a score ranging from 0-4. In total, the lowest 0 and the highest 36 points can be obtained. High scores indicate low back awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- HAZAL genç, Istanbul, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No